CLINICAL TRIAL: NCT03231969
Title: A Single-Center, Double-Masked, Randomized, Vehicle-Controlled, Phase 2, Dose Ranging Evaluation of the Effectiveness of Bilastine Ophthalmic Solution (0.2%, 0.4%, and 0.6%) Compared to Vehicle for the Treatment of Allergic Conjunctivitis in the Conjunctival Allergen Challenge (Ora-CAC®) Model
Brief Title: A Single-Center, Phase 2 Study Evaluating Bilastine Ophthalmic Solution in the CAC® Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BOFT-0117/DR-CAC
Record Dates: First submitted 2017-07-20; First posted 2017-07-27 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2021-10

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Bilastine 0.2% (Experimental): Bilastine Ophthalmic solution 0.2%
  1 drop in each eye at 3 separate times during a 25 day period.
  Interventions: Drug: Bilastine 0.2%
- Bilastine 0.4% (Experimental): Bilastine Ophthalmic solution 0.4%
  1 drop in each eye at 3 separate times during a 25 day period.
  Interventions: Drug: Bilastine 0.4%
- Bilastine 0.6% (Experimental): Bilastine Ophthalmic solution 0.6%
  1 drop in each eye at 3 separate times during a 25 day period.
  Interventions: Drug: Bilastine 0.6%
- Bilastine 0% (Placebo Comparator): Vehicle of Bilastine Ophthalmic Solution
  1 drop in each eye at 3 separate times during a 25 day period.
  Interventions: Drug: Bilastine 0%

INTERVENTIONS:
Drug: Bilastine 0.2% — 1 drop in each eye at 3 separate times during a 25 day period.
  Arms: Bilastine 0.2%
Drug: Bilastine 0.4% — 1 drop in each eye at 3 separate times during a 25 day period.
  Arms: Bilastine 0.4%
Drug: Bilastine 0.6% — 1 drop in each eye at 3 separate times during a 25 day period.
  Arms: Bilastine 0.6%
Drug: Bilastine 0% — 1 drop in each eye at 3 separate times during a 25 day period.
  Arms: Bilastine 0%

SUMMARY:
To evaluate the efficacy of Bilastine Ophthalmic Solution (0.2%,0.4%,0.6%) compared to vehicle for the treatment of the signs and symptoms of allergic conjunctivitis

ELIGIBILITY:
Key Inclusion Criteria:

* be at least 18 years old
* be willing and able to avoid all disallowed medications and contact lenses
* must have a pregnancy test if of childbearing potential
* must be able to read an eye chart from 10 feet away

Key Exclusion Criteria:

* must not have any allergies to the study medications
* must not have any ocular or non ocular condition that investigator feels will interfere with study parameters
* must not have used immunotherapy in the last 2 years
* must not have used an investigational drug or device in the past 30 days or concurrently enrolled in another investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ora Clinical Research Center, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bilastine 0.2% | Bilastine 0.4% | Bilastine 0.6% | Bilastine 0%
Started | 30 | 30 | 31 | 30
Completed | 28 | 28 | 30 | 30
Not Completed | 2 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilastine 0.2% | Bilastine 0.4% | Bilastine 0.6% | Bilastine 0% | Total
Number analyzed (Participants) | 30 | 30 | 31 | 30 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 27 | 27 | 109
  >=65 years | 2 | 3 | 4 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (10.7) | 47.0 (13.95) | 51.8 (13.4) | 48.3 (13.24) | 49.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 15 | 17 | 66
  Male | 14 | 12 | 16 | 13 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 4 | 5 | 19
  Not Hispanic or Latino | 27 | 23 | 27 | 25 | 102
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 4 | 3 | 10
  White | 27 | 27 | 26 | 27 | 107
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 31 | 30 | 121
Ocular Itching- Baseline [Mean (Standard Deviation); unit: units on a scale] — The primary efficacy measure was ocular itching evaluated by the subject post-CAC at Visit 4b (Day 1, 16h post treatment), Visit 5b (Day 15 ±3, 8h post treatment), and Visit 6 (Day 22 ±3, 15 minutes post treatment), using a 0 to 4 Ora Calibra scale: 0 = none (normal, no itching), 4 = incapacitating itch.The baseline measures for this primary outcome will be the "pre-CAC" values (pre-Conjunctival Allergen Challenge).
  units on a scale
    Visit 4b: Pre- CAC | 0.058 (0.2043) | 0.000 (0.0000) | 0.048 (0.1981) | 0.025 (0.1006) | 0.03275 (0.12575)
    Visit 5b: Pre- CAC | 0.000 (0.0000) | 0.000 (0.0000) | 0.033 (0.1826) | 0.033 (0.1826) | 0.0165 (0.0913)
    Visit 6: Pre- CAC | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: The primary efficacy measure was ocular itching evaluated by the subject post-CAC (Conjunctival Allergen Challenge) at Visits 4b, 5b, and 6, using a 0 to 4 Ora Calibra scale: 0 = none (normal, no itching), 4 = incapacitating itch.
Time Frame: The outcome measure was assessed at Visit 4b (Day 1, 16h post treatment), Visit 5b (Day 15 ±3, 8h post treatment), and Visit 6 (Day 22 ±3, 15 minutes post treatment).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Bilastine 0% (Vehicle): Bilastine 0%: 1 drop in each eye at 3 separate times during a 25 day period
Arm/Group | Bilastine 0.2% | Bilastine 0.4% | Bilastine 0.6% | Bilastine 0% (Vehicle)
Number analyzed (Participants) | 30 | 30 | 31 | 30
units on a scale
  Visit 4b: 3 minutes Post-CAC | 1.908 (0.7809) | 1.925 (0.9449) | 1.177 (1.0332) | 2.758 (0.7146)
  Visit 4b: 5 minutes Post-CAC | 2.075 (0.7828) | 2.117 (0.9531) | 1.218 (1.1268) | 3.017 (0.5979)
  Visit 4b: 7 minutes Post-CAC | 2.092 (0.7698) | 2.100 (1.0760) | 1.218 (1.1157) | 2.917 (0.5884)
  Visit 5b: 3 minutes Post-CAC | 1.397 (1.1050) | 1.250 (0.8872) | 0.708 (0.8908) | 2.558 (0.8032)
  Visit 5b: 5 minutes Post-CAC | 1.466 (0.9300) | 1.464 (0.9592) | 0.817 (1.0503) | 2.642 (0.7505)
  Visit 5b: 7 minutes Post-CAC | 1.379 (0.8573) | 1.518 (1.0340) | 0.742 (0.9837) | 2.642 (0.7704)
  Visit 6: 3 minutes Post-CAC | 0.679 (0.6662) | 0.732 (0.9127) | 0.392 (0.5749) | 2.542 (0.8384)
  Visit 6: 5 minutes Post-CAC | 0.920 (0.7235) | 1.143 (0.9987) | 0.558 (0.6355) | 2.592 (0.8343)
  Visit 6: 7 minutes Post-CAC | 1.000 (0.7454) | 1.214 (0.9421) | 0.583 (0.6706) | 2.483 (0.9024)
Statistical Analysis 1: Comparison: Bilastine 0.2% vs Bilastine 0% (Vehicle); Treatment difference (95%CI): Bilastine 0.2% arm minus Bilastine 0% (Vehicle) arm at Visit 4b (including all time points); Test type: Superiority; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -0.791, 95% CI 2-sided [-1.203 to -0.378]
Statistical Analysis 2: Comparison: Bilastine 0.4% vs Bilastine 0% (Vehicle); Treatment difference (95%CI): Bilastine 0.4% arm minus Bilastine 0% (Vehicle) arm at Visit 4b (including all time points); Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -0.851, 95% CI 2-sided [-1.263 to -0.439]
Statistical Analysis 3: Comparison: Bilastine 0.6% vs Bilastine 0% (Vehicle); Treatment difference (95%CI): Bilastine 0.6% arm minus Bilastine 0% (Vehicle) arm at Visit 4b (including all time points); Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -1.545, 95% CI 2-sided [-1.954 to -1.135]
Statistical Analysis 4: Comparison: Bilastine 0.2% vs Bilastine 0% (Vehicle); Treatment difference (95%CI): Bilastine 0.2% arm minus Bilastine 0% (Vehicle) arm at Visit 5b (including all time points); Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -1.208, 95% CI 2-sided [-1.639 to -0.778]
Statistical Analysis 5: Comparison: Bilastine 0.4% vs Bilastine 0% (Vehicle); Treatment difference (95%CI): Bilastine 0.4% arm minus Bilastine 0% (Vehicle) arm at Visit 5b (including all time points); Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -1.245, 95% CI 2-sided [-1.679 to -0.811]
Statistical Analysis 6: Comparison: Bilastine 0.6% vs Bilastine 0% (Vehicle); Treatment difference (95%CI): Bilastine 0.6% arm minus Bilastine 0% (Vehicle) arm at Visit 5b (including all time points); Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -1.846, 95% CI 2-sided [-2.273 to -1.418]
Statistical Analysis 7: Comparison: Bilastine 0.2% vs Bilastine 0% (Vehicle); Treatment difference (95%CI): Bilastine 0.2% arm minus Bilastine 0% (Vehicle) arm at Visit 6 (including all time points); Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -1.696, 95% CI 2-sided [-2.080 to -1.312]
Statistical Analysis 8: Comparison: Bilastine 0.4% vs Bilastine 0% (Vehicle); Treatment difference (95%CI): Bilastine 0.4% arm minus Bilastine 0% (Vehicle) arm at Visit 6 (including all time points); Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -1.617, 95% CI 2-sided [-2.001 to -1.232]
Statistical Analysis 9: Comparison: Bilastine 0.6% vs Bilastine 0% (Vehicle); Treatment difference (95%CI): Bilastine 0.6% arm minus Bilastine 0% (Vehicle) arm at Visit 6 (including all time points); Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -2.009, 95% CI 2-sided [-2.387 to -1.630]

ADVERSE EVENTS:
Time Frame: Safety assessment period (Day 1 through Day 22). Adverts events were assessed at all office visits, throughout a period of 22 days.
Arm/Group | Bilastine 0.2% | Bilastine 0.4% | Bilastine 0.6% | Bilastine 0%
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 8/30 | 3/30 | 1/31 | 7/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bilastine 0.2% (N=30) | Bilastine 0.4% (N=30) | Bilastine 0.6% (N=31) | Bilastine 0% (N=30)
Visual Acuity Reduced (Eye disorders) | 2 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0
Corneal Deposits (Eye disorders) | 0 | 0 | 0 | 1
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 1 | 0 | 0
Macular Fibrosis (Eye disorders) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 3
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03231969/Prot_SAP_001.pdf